CLINICAL TRIAL: NCT02961231
Title: Evaluation of PCV Schedules in a Naive Population in Vietnam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nagasaki University (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); Murdoch Childrens Research Institute (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Prof.Lay-Myint Yoshida, Professor, Department of Pediaric Infectious Diseases, Institute of Tropical Medicine, Nagasaki University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPP1139859
Record Dates: First submitted 2016-11-01; First posted 2016-11-10 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pneumonia, Pneumococcal
Keywords: Pneumococcal conjugate vaccine; Herd immunity; Reduced dosing schedule
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — PHiD-CV vaccine

STUDY DESIGN:
Masking Description: 43068 children participated in the PCV vaccination activity during the study period.
  A total of 18652 children were enrolled in the pneumococcal carriage surveys to evaluate the non-inferiority of VT reduction in 1p+1, 0p+1 vs 2p+1 and 3p+0 arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (4):
- PCV 2p+1 (Active Comparator): PCV 2p+1 schedule: WHO recommended 2 primary at 2, 4 months and a booster dose at 12 month
  Interventions: Biological: PCV 2p+1
- PCV 3p+0 (Active Comparator): PCV 3p+0 schedule: WHO recommended 3 primary doses at 2, 3 and 4 months
  Interventions: Biological: PCV 3p+0
- PCV 1p+1 (Experimental): PCV 1p+1 schedule: one primary dose at 2 month and a booster at 12 month
  Interventions: Biological: PCV 1p+1
- PCV 0p+1 (Experimental): PCV 0p+1 schedule: no primary dose, only a booster at 12 month
  Interventions: Biological: PCV 0p+1

INTERVENTIONS:
Biological: PCV 2p+1 — introduction of PCV in a reduced dosing 2p+1 schedule
  Other Names: Synflorix
  Arms: PCV 2p+1
Biological: PCV 3p+0 — introduction of PCV in a reduced dosing 3p+0 schedule
  Other Names: Synflorix
  Arms: PCV 3p+0
Biological: PCV 1p+1 — introduction of PCV in a reduced dosing 1p+1 schedule
  Other Names: Synflorix
  Arms: PCV 1p+1
Biological: PCV 0p+1 — introduction of PCV in a reduced dosing 0p+1 schedule
  Other Names: Synflorix
  Arms: PCV 0p+1

SUMMARY:
The cost of pneumococcal conjugate vaccine use can be greatly reduced by making use of existing herd immunity to protect children against vaccine type pneumococci. The investigators will reduce the circulation of vaccine type pneumococci to low levels by PCV catch-up campaign; vaccinating all children less than 3 years of age with PCV, after which the investigators will evaluate the ability of a simplified two doses regimen and an alternative one dose regimen to prevent the reintroduction of vaccine type pneumococci compared to the WHO recommended 2 doses schedule.

DETAILED DESCRIPTION:
Background Pneumococcal conjugate vaccine (PCVs) have substantially reduced the burden of pneumococcal disease. WHO currently recommends giving PCVs as 3 doses - either 3 doses in infancy with Pentavalent vaccine (3p+0), or two doses in infancy followed by a booster around the end of the first year of life (2p+1). The 3p+0 schedule is used in many countries introducing PCV with Gavi support while several European countries are using 2p+1 schedule. However, their high price and the current recommendation for at least 3 doses to achieve full individual protection for infants, introduces a substantial financial burden. As a result, many middle income countries have not yet introduced PCVs, and low income countries that have introduced PCVs with the aid of the Gavi, the Vaccine Alliance, may not be able to sustain PCV vaccination after graduating from GAVI support.

To date PCV programs have been designed to provide optimal individual protection of the vaccinees, yet experience in developed countries indicates that herd immunity, which is generated by reducing carriage and hence transmission of vaccine serotypes in the community, controls vaccine type pneumococcal disease in vaccinated and unvaccinated individuals alike [1]. Using PCV impact on vaccine type carriage as a marker of vaccine type disease [2], the investigators will investigate the feasibility of reducing the number of infant doses in the PCV immunization schedule, to make more efficient use of herd immunity in the protection against pneumococcal disease.

Study aim and objectives Primary objective 1- The investigators will measure the effect of the 1p+1 schedule on vaccine type pneumococcal carriage and non-inferiority compared to a 2p+1 or 3p+0 schedule in (a) children aged 4-11 months, i.e. after the age of a completed primary series and before the age where they would receive a booster dose (this is the population that is most at risk for pneumococcal disease and is likely to receive less direct protection from a reduced primary series), and (b) children aged 14-24 months, i.e. after the age where a booster dose is given in the treatment arms(this is the beginning of the age period when most intense transmission of pneumococci is believed to occur).

Secondary objective 1 - The investigators will measure the effect (both direct + indirect effects) of the 0p+1 schedule against vaccine type carriage and non-inferiority against a 2p+1 or/and 3p+0 schedules respectively in (a) children aged 4-11 months, and (b) children aged 14-24 months,.

Secondary objective 2 - The investigators will measure the effect of the 1p+1 and 0p+1 schedules against vaccine type carriage and non-inferiority against a 2p+1 or 3p+0 schedules respectively among unvaccinated mothers.

Secondary Objective 3- The investigators will measure the effect of catchup vaccination effect in the community by conducting and post catchup carriage survey, 4 months after the second catchup vaccination campaign.

Secondary objective 4 - The investigators will develop mathematical models to predict the impact of 1p+1 and 0p+1 schedules against vaccine type carriage and disease in Nha Trang if introduced simultaneously to all clusters following a catch up campaign, and infer the impact of such schedules in other transmission settings.

Study site: The study will be conducted in 27 communes of Nha Trang, central Vietnam which is the capital of Khánh Hòa province and has about 400,000 inhabitants. PCV10 was recently registered in Vietnam. However, PCV is yet to be introduced into the national immunization program in Vietnam.

Study design: The investigators will conduct a PCV cluster randomized trial in 27 communes of Nha Trang city. There will be four different schedules of PCV intervention arms; 1p+1, 0p+1, 2p+1, and 3p+0 schedules. The followings are the PCV schedules that will be investigate in this study.

0p+1 - A single dose of PCV at 12 months of age

1. p+1 - A two-dose schedule of PCV at 2 and 12 months of age
2. p+1 - A three-dose schedule of PCV at 2, 4 and 12 months of age
3. p+0 - A three dose schedule of PCV at 2, 3 and 4 months of age Communes will be considered as clusters. Six clusters for each intervention arm and 3 clusters for the unvaccinated arm will be included in the study.

Selection of PCV for the study: PCV10 has recently been registered in Vietnam and can be purchased locally, while this is not yet the case for PCV13. Therefore the investigators decided to use PCV10 for the study.

Pneumococcal carriage survey: Nasopharyngeal samples will be collected before the catchup vaccination and annually from 60 subjects per age groups (4-11mth, 14-24mth) and their mothers. The investigators will include 6 clusters for each intervention arm. Sixty subjects will be recruited from 3 age groups (60 children 4 to 11 months old, 60 children 14 to 24 months old and 120 mothers) of each clusters to achieve the primary study objectives, which accumulates to 6480 samples for each cross sectional pneumococcal carriage survey. Our carriage surveys in Nha Trang among healthy children as well as hospitalized children admitted with acute respiratory infection found similar serotype coverage for both PCV10 and PCV13 (~65% in health and ~70% in ARI children respectively)[3]. Number of cluster and sample size were calculated based on Hayes and Moulton [4].

Selection of intervention communes: The 3 communes in the north; Vinh Luong, Vinh Phuong, and Vinh Hoa will be selected as unvaccinated communes based on the geographical background. Although we will not consider these communes as controls for the study, inclusion of unvaccinated communes will provide information on potential year by year carriage due to introduction of new strains from outside of Nha Trang or from vaccinated communes in Nha Trang. The remaining 24 communes will be randomized into 4 arms: a 2p+1 arm, a 3p+0 arm, a 1p+1 arm, and a 0p+1 arm. There are 8 rural and 19 urban communes in Nha Trang City. Two rural communes and one urban commune were selected for the unvaccinated cluster so there were 6 rural and 18 urban communes left for the randomization.

Initial catchup vaccination: a catch up vaccination campaign will be done before the start of PCV vaccine introduction. Three doses of PCV10 will be administered to all children between 2 - 6 months of age with an interval of 2 months between the first and second, and 7 months between the second and the third doses. A catch up of two doses of PCV10 will be administered to all children between 7 and 18 months of age with an interval of two months between the two doses. Children between 19 and 36 months of age will receive a single dose. This is expected to quickly control circulation of vaccine serotypes in these areas. The total number of children less than 3 years of age in 24 communes is estimated to be approximately 18,000 (750 x 24). The total number of vaccine doses required is estimated to be 30,000 doses.

PCV introduction in birth cohort children: There will be 4 PCV intervention schedules; 2p+1 arm, 3p+0 arm, 1p+1 arm, and 0p+1 arm in this study. The children will receive PCV based on which cluster/communes they reside in. This PCV vaccination work will start one month after the initial catchup vaccination campaign. Based on the current census data, the investigators estimate that the birth cohort of children in each communes will be 250 and there will be a total of 6000 children to be vaccinated per year in 24 treatment communes. Vietnam National Immunization Program vaccinate DPT-HepB-Hib vaccine at 2, 3, 4months and JE vaccine at 12 months. The investigators will vaccinate PCV on the same visit with the above vaccines.

Sample collection and testing: Nasopharyngeal samples will be collected from the study subjects. The initial screening test will be conducted at Nha Trang Pasteur Institute. DNA will be extracted from the nasopharyngeal samples and screened for S.pneumoniae lytA gene by realtime PCR assay. The positive samples will be cultured, DNA extracted and then the DNA samples will be transported to MCRI for serotype determination by Microarray assay. Already standardized protocols will be used for the testing [5].

Approach and data analysis: To address primary objective and secondary objective 1, 2 & 3 we will conduct annual cross sectional nasopharyngeal carriage surveys testing 60 children 4 to 11 months old, 60 children 14 to 24 months old and their mothers in each cluster for the presence of vaccine serotype carriage in 27 communes of Nha Trang. The comparison of the baseline and post-catchup vaccination carriage survey will reveal the effect of catchup vaccination to children <3 years of age and initial vaccination in the community. The comparison of carriage prevalence in the intervention/treatment (1p+1 or 0p+1) clusters and the gold standard (2p+1 or 3p+0) clusters respectively will allow age-group specific assessment of non-inferiority of the 1p+1 and 0p+1 schedules if compared with the 2p+1 or 3p+0 schedules respectively in regard to protection against vaccine type carriage.

Mathematical modelling analysis: Furthermore we will use the acquired data to fit a dynamic metapopulation model for pneumococcal transmission to the observed changes in pneumococcal carriage in the 27 study communes. The estimated model parameters will be used to predict the impact of PCV in a scenario where PCV had been introduced using the 1p+1 or 0p+1 schedules in all 27 communes. We will also use this framework to infer the impact of continuation with a 1p+1 or 0p+1 schedules in other transmission settings where PCVs have been in use and where high quality allows model calibration (secondary objective 4).

Severe adverse events monitoring: Preventive medicine center in Nha Trang is responsible for monitoring SAE/AE related to routine national vaccination program in Nha Trang will collaborate and support on PCV related SAE monitoring activities.

Timeline: The investigators have already received ethical approval from Nagasaki University, Nagasaki and National Institute of Hygiene and Epidemiology, Hanoi. Ministry of Health, Vietnam approval was also obtained in September 2016.

2016, October: Initial carriage study, followed by yearly carriage surveys at same month every year up to 5 years.

2017 February: First catch-up vaccination (the second and third catch-up vaccination will follow 2 months after the first dose and 7 months after the second dose) 2017 March: Start the PCV introduction in 24 communes with different schedule based on their cluster allocation. This PCV introduction will be for 5 years.

2017, June: Post-catchup carriage survey Annual cross sectional carriage surveys will be conducted in the same month with the baseline carriage survey in 2017, 2018, 2019, 2020 and 2021 respectively.

ELIGIBILITY:
Inclusion Criteria: All children living in the intervention communes in Nha Trang city, whose parents or guardian give informed consent will be eligible to receive PCV in accordance with their age.

Exclusion Criteria: Children who are not fit enough to receive national vaccination program vaccine for health reason (eg.fever, currently under medication due to illness such as pneumonia, diarrhea, etc) in accordance with Vietnam national immunization guidelines. This will be decided by the medical doctor in charge of the vaccination at commune health center in accordance with Vietnamese guideline.

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18652 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
vaccine type pneumococcal carriage | up to 60 months after PCV intervention
  Vaccine type pneumococcal carriage among children receiving different PCV dose will be investigated yearly. Non-inferiority of 1p+1 dose will be compared with those receiving 2p+1/3p+0 groups.

CONTACTS AND LOCATIONS:
Overall Officials: LAYMYINT YOSHIDA, MBBS, PhD, Principal Investigator — Institute of Tropical Medicine, Nagasaki University, Nagasaki
Locations (1):
- Commune Health Centers, Nha Trang, Khanh Hoa, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] R. J. Hayes, L. H. Moulton, Cluster randomised trials (Chapman & Hall, 2009).
- [Background] Satzke C, Dunne EM, Porter BD, Klugman KP, Mulholland EK; PneuCarriage project group. The PneuCarriage Project: A Multi-Centre Comparative Study to Identify the Best Serotyping Methods for Examining Pneumococcal Carriage in Vaccine Evaluation Studies. PLoS Med. 2015 Nov 17;12(11):e1001903; discussion e1001903. doi: 10.1371/journal.pmed.1001903. eCollection 2015 Nov. PMID 26575033
- [Result] Bogaert D, De Groot R, Hermans PW. Streptococcus pneumoniae colonisation: the key to pneumococcal disease. Lancet Infect Dis. 2004 Mar;4(3):144-54. doi: 10.1016/S1473-3099(04)00938-7. PMID 14998500
- [Result] Feikin DR, Kagucia EW, Loo JD, Link-Gelles R, Puhan MA, Cherian T, Levine OS, Whitney CG, O'Brien KL, Moore MR; Serotype Replacement Study Group. Serotype-specific changes in invasive pneumococcal disease after pneumococcal conjugate vaccine introduction: a pooled analysis of multiple surveillance sites. PLoS Med. 2013;10(9):e1001517. doi: 10.1371/journal.pmed.1001517. Epub 2013 Sep 24. PMID 24086113
- [Result] Vu HT, Yoshida LM, Suzuki M, Nguyen HA, Nguyen CD, Nguyen AT, Oishi K, Yamamoto T, Watanabe K, Vu TD. Association between nasopharyngeal load of Streptococcus pneumoniae, viral coinfection, and radiologically confirmed pneumonia in Vietnamese children. Pediatr Infect Dis J. 2011 Jan;30(1):11-8. doi: 10.1097/INF.0b013e3181f111a2. PMID 20686433
- [Derived] Yoshida LM, Toizumi M, Nguyen HAT, Quilty BJ, Lien LT, Hoang LH, Iwasaki C, Takegata M, Kitamura N, Nation ML, Hinds J, van Zandvoort K, Ortika BD, Dunne EM, Satzke C, Do HT, Mulholland K, Flasche S, Dang DA. Effect of a Reduced PCV10 Dose Schedule on Pneumococcal Carriage in Vietnam. N Engl J Med. 2024 Nov 28;391(21):1992-2002. doi: 10.1056/NEJMoa2400007. PMID 39602629
- [Derived] Yoshida LM, Flasche S, Mulholland K, Nguyen HA, Nguyen C, Toizumi M, Dang DA. Evaluation of the effect of reduced-dose pneumococcal conjugate vaccine schedules on vaccine serotype carriage in children and their caretakers in a naive population in Vietnam: Protocol for a cluster randomized non-inferiority trial. Gates Open Res. 2023 Jul 20;7:110. doi: 10.12688/gatesopenres.14742.1. eCollection 2023. PMID 37780234